CLINICAL TRIAL: NCT07044310
Title: Phase 2 Trial of 5-Strain Probiotic Formulation in Hormone Receptor-Positive Breast Cancer Receiving Aromatase Inhibitor to Prevent Bone Loss
Brief Title: 5-strain Probiotic Formulation in HR-positive Breast Cancer Receiving Aromatase Inhibitor to Prevent Bone Loss
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC240302; NCI-2025-04267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-007055 (Other: Mayo Clinic Institutional Review Board); MC240302 (Other: Mayo Clinic)
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Specimen Handling; Bone Density; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (WBF-038) (Experimental): Patients receive WBF-038 PO QD for 365 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and BMD test at screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Mineral Density Test; Other: Questionnaire Administration; Drug: WBF-038

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Mineral Density Test — Undergo BMD
  Other Names: BMD; bone density; Bone Density Test; bone mass; Bone Mineral Density
Other: Questionnaire Administration — Ancillary studies
Drug: WBF-038 — Given WBF-038 PO
  Other Names: Akkermansia muciniphila/Anaerobutyricum hallii/Bifidobacterium infantis/Clostridium beijerinckii/Clostridium butyricum/Inulin WBF-038; Pendulum WBF-038 (SY); Probiotic/Prebiotic Formulation WBF-038 (SY); Synbiotic Formulation WBF-038 (SY); WBF 038 (CN); WBF-038 (CN); WBF038 (CN)

SUMMARY:
This phase II trial tests how well a probiotic, WBF-038, works in preventing bone loss in patients with early-stage hormone receptor-positive breast cancer who are starting treatment with aromatase inhibitors. Aromatase inhibitors are a drug that blocks the activity of an enzyme called aromatase, which the body uses to make estrogen in the ovaries and other tissues. Blocking aromatase lowers the amount of estrogen made by the body, which may stop the growth of cancer cells that need estrogen to grow. Aromatase inhibitors are used to treat some types of breast cancer or to keep it from coming back. Aromatase inhibitors can affect bone health, weight, blood sugar, and waist size. WBF-038 is a combination of both prebiotics and probiotics, designed to improve metabolic health. Giving WBF-038 may improve bone turnover, bone health, blood sugar, weight, and waist circumference in patients with early-stage hormone receptor-positive breast cancer starting on adjuvant endocrine therapy with an aromatase inhibitor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the median percent change from baseline (prior to the start of an aromatase inhibitor [AI]) at 15 months in C-terminal telopeptide of type 1 collagen (CTx) in early-stage breast cancer patients who receive WBF-038 treatment for 12 months starting at 3 months post-baseline.

SECONDARY OBJECTIVES:

I. To evaluate the median percent change from baseline (prior to the start of an AI) at 15 months in the lumbar spine and hip bone mineral density in early-stage breast cancer patients who receive WBF-038 treatment for 12 months starting at 3 months post-baseline.

II. To evaluate safety and risk of fracture associated with WBF-038.

EXPLORATORY OBJECTIVES:

I. To evaluate changes from baseline (prior to the start of an AI) over time in CTx, alkaline phosphatase (ALK), fasting blood sugar (FBS), hemoglobin A1C (HbA1C), and Procollagen I Intact N-Terminal (P1NP) at 3, 6, 15, and 18 months post-baseline.

II. To evaluate changes from baseline (prior to the start of an AI) over time in weight and waist circumference at 3, 6, 15, and 18 months post-baseline.

III. To evaluate changes in the cytokine profile over time. IV. To evaluate the association between stool microbiome, stool short-chain fatty acid (SCFA), and serum SCFA and changes over time in CTx and lumbar spine and hip bone mineral density.

V. To evaluate changes over time in AI-associated musculoskeletal symptoms (AIMSS) with patient-reported outcomes (PRO) using the Stanford Health Assessment Questionnaire (HAQ) and pain visual analog scale (VAS).

OUTLINE:

Patients receive WBF-038 orally (PO) once daily (QD) for 365 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and bone mineral density (BMD) test at screening and on study.

After completion of study intervention, patients are followed up at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Histologically confirmed anatomical stage 0-III hormone receptor-positive breast cancer
* Will be starting on an aromatase inhibitor (letrozole, anastrozole, or exemestane) ± ovarian function suppression (OFS) per treating physician's discretion
* Absolute neutrophil count (ANC) ≥ 1000/mm^3 (prior to registration)
* Platelet count ≥ 75,000/mm^3 (prior to registration)
* Hemoglobin ≥ 9.0 g/dL (prior to registration)
* Creatinine ≤ 2 x upper limit of normal (ULN) (prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) ≤ 2 x ULN (prior to registration)
* Albumin ≥ 3 g/dL (prior to registration)
* Willing and able to provide research stool and blood samples
* Negative serum pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only (< 60 years old with intact uterus)
* Capable of providing valid informed consent
* Willing to return to enrolling institution for all study visits (blood draws, etc)

Exclusion Criteria:

* Requires prolonged systemic antibiotic therapy for other conditions and recent systemic antibiotic ≤ 14 days prior to registration
* Fecal microbiota transplant (FMT) ≤ 6 months prior to registration
* FMT with an associated serious adverse event related to the FMT product or procedure
* Co-morbid systemic illnesses or other severe concurrent diseases which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of over-the-counter probiotics
* Immunocompromised patients including patients known to be HIV positive or those on chronic steroids > 20 mg prednisone a day or prednisone-equivalent. Note: Must be off systemic steroids ≥ 90 days prior to registration. However, topical steroids, inhalants, or steroid eye drops are permitted
* History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis
* History of chronic diarrhea
* History of celiac disease
* Currently has a colostomy
* Intraabdominal surgery related to gastrointestinal tract ≤ 60 days prior to registration
* Evidence of active, severe colitis
* History of short gut syndrome or motility disorders
* Requires the daily use of medications to manage bowel hypermotility, such as imodium or lomotil
* Active autoimmune disease that has required systemic treatment in the ≤ 30 days (i.e., with the use of disease-modifying agents, corticosteroids, or immunosuppressive products) prior to registration. Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment ≤ 30 days prior to registration are not excluded
* History of osteoporosis or hyperparathyroidism
* History of untreated vitamin D deficiency
* Receiving or will receive bisphosphonates during study period (alendronate, risedronate, ibandronate, pamidronate, or zolendronic acid) or denosumab
* Patients who received oral bisphosphonate within ≤ 12 weeks, intravenous (IV) zoledronic acid (Reclast) ≤ 52 weeks, or denosumab ≤ 24 weeks will also be excluded
* Known hypersensitivity to any component of study product (including known inulin intolerance)
* Known hypersensitivity to > 4 first-line antimicrobial therapies against akkermansia muciniphila, clostridium beijerinckii, clostridium butyricum, anaerobutyricum hallii, including penicillin, piperacillin, tetracycline, amoxicillin, or ampicillin
* Known hypersensitivity to > 4 first line antimicrobial therapies against bifidobacterium infantis Bi-26TM, including gentamicin, kanamycin, streptomycin, tetracycline, erythromycin, clindamycin, ampicillin, vancomycin
* Received an experimental product ≤ 30 days prior to registration
* Receiving or will receive CDK 4/6 inhibitor (abemaciclib, ribociclib, or palbociclib)
* Received chemotherapy ≤ 30 days prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in C-terminal telopeptide of type 1 collagen (CTx) | Baseline; 90 days after start of AI therapy (before beginning WBF-038); 14 days after start of WBF-038; 90 days after start of WBF-038; 180 days after start of WBF-038; 365 days after start of WBF-038; 90 days after stopping WBF-038
  Assessed by standard lab tests at baseline (at study enrollment/eligibility assessment before any therapy) followed by 6 study visits. Participants receive aromatase Inhibitor (AI) therapy followed by a one-year course of probiotic WBF-038.

SECONDARY OUTCOMES:
Change in lumbar spine mineral density | Baseline; 365 days after start of WBF-038
  Will be measured by central dual energy x-ray absorptiometry. Participants receive aromatase Inhibitor (AI) therapy followed by a one-year course of probiotic WBF-038.
Change in hip bone mineral density | Baseline; 365 days after start of WBF-038
  Will be measured by central dual energy x-ray absorptiometry. Participants receive aromatase Inhibitor (AI) therapy followed by a one-year course of probiotic WBF-038.
Incidence of adverse events | Baseline; 90 days after start of AI therapy (before beginning WBF-038); 90 days after start of WBF-038; 365 days after starting WBF-038; 90 days after stopping WBF-038;
  Will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials